CLINICAL TRIAL: NCT07230717
Title: Clinical and Radiographic Evaluation of Pulpotomy Versus Pulpectomy in Primary Molars With Irreversible Pulpitis or Necrotic Pulp: A Split-Mouth Randomized Clinical Trial
Brief Title: Evaluation of Pulpotomy Versus Pulpectomy in Primary Molars With Irreversible Pulpitis or Necrotic Pulp
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ajman University (Other)
Responsible Party: Principal Investigator, Dr. Raghavendra Shetty, Associate Professor, Ajman University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D-S-H-22-Jun
Record Dates: First submitted 2025-09-17; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pulp Therapy; Pulpitis - Irreversible; Pulp Necrosis
Keywords: Pulpotomy; Pulpectomy; primary molars; irreversible pulpitis; necrotic pulp
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Pulpotomy; Pulpectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulpotomy (Experimental): Pulpotomy
  Interventions: Procedure: Pulpotomy
- Pulpectomy (Active Comparator): Pulpectomy
  Interventions: Procedure: Pulpectomy

INTERVENTIONS:
Procedure: Pulpotomy — Pulpotomy with pulpotec Powder: (iodoform, polyoxymethylene, excipient) and a Liquid: (dexamethasone acetate, formaldehyde, phenol, guaiacol, excipient) mixed into a paste consistency as per manufacturer instruction.
  Pulpectomy with metapex Content: Calcium Hydroxide, Iodoform, Silicon oil
  Arms: Pulpotomy
Procedure: Pulpectomy — Calcium Hydroxide, Iodoform, Silicon oil
  Arms: Pulpectomy

SUMMARY:
Preserving primary teeth until their normal exfoliation time is crucial for maintaining the child's normal function, esthetics, arch integrity, and correct eruption of permanent successors. Given the growing interest in conservative procedures and the clinical need for simpler, more predictable pulp therapy outcomes in children, evaluating pulpotomy with Pulpotec as a potential alternative to pulpectomy is essential.

The aim of this study is to evaluate the clinical and radiographic success of pulpotomy using Pulpotec versus pulpectomy using Metapex, a calcium hydroxide with iodoform paste, to treat primary molars in children diagnosed with irreversible pulpitis or necrotic pulp in the Postgraduate Pediatric Dental Clinic at Ajman University, UAE. A total of 25 contralateral paired molar samples from children aged 4 to 8 will be included in this split-mouth randomized controlled study. Each child will serve as their own control, with one tooth randomized to the intervention group (Pulpotomy using Pulpotec) and the other to the control group (Pulpectomy using Metapex) to assess patients' clinical and radiographic outcomes over a 12-month follow-up period. Patients will have their dental anxiety psychometrically assessed using the RMS pictorial scale. In addition, a pulse oximeter will be used as a biological marker in the study to measure oxygen saturation and pulse rate.

DETAILED DESCRIPTION:
With increasing emphasis on conservative and predictable pulp therapy in pediatric dentistry, this study aims to evaluate pulpotomy using Pulpotec as a potential alternative to pulpectomy using Metapex in the management of primary molars with irreversible pulpitis or necrotic pulp.

This split-mouth randomized controlled clinical trial will include 25 children aged 4-8 years attending the Postgraduate Pediatric Dental Clinic at Ajman University, UAE. Each participant will contribute two contralateral primary molars-one assigned to the intervention group (Pulpotomy with Pulpotec) and the other to the control group (Pulpectomy with Metapex, a calcium hydroxide and iodoform paste).

The outcome will assess and compare the clinical and radiographic success rates of pulpotomy and pulpectomy procedures performed in primary molars diagnosed with irreversible pulpitis or necrotic pulp. Clinical success will be defined by the absence of pain, swelling, sinus tract, mobility, or tenderness to percussion. Radiographic success will be defined by the absence of periapical or inter-radicular radiolucency, internal or external resorption, and evidence of continued root resorption consistent with normal exfoliation. In addition, dental anxiety will be assessed using the RMS Pictorial Anxiety Scale, and physiological parameters such as pulse rate (beats/min) and oxygen saturation (SpO₂, %) will be recorded using a pulse oximeter to explore potential correlations between anxiety and treatment response.

ELIGIBILITY:
Inclusion Criteria

* Patients in healthy medical conditions
* Bilateral/contralateral primary molars diagnosed with irreversible pulpitis or necrotic pulp
* Periapical or bifurcation radiolucency
* Chronic apical intraoral abscess
* Sinus tract or fistula formation
* No tooth mobility or grade I mobility
* External root resorption less than or equal to 1/3rd of the roots
* Tooth should be restorable

Exclusion Criteria

* Patients who are medically compromised (with systemic conditions)
* Acute extraoral abscess
* Grade II or III tooth mobility
* External root resorption in more than 1/3 of roots
* Physiological root resorption of more than 1/3 of the roots or near exfoliation
* Non-restorable teeth

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiographic success rates of pulpotomy versus pulpectomy in primary molars of children with irreversible pulpitis or necrotic pulp over a 12-month follow-up period | 3 months, 6 months, 9 months, and 12 months follow up post-treatment.
  The outcome will assess and compare the clinical and radiographic success rates of pulpotomy and pulpectomy procedures performed in primary molars diagnosed with irreversible pulpitis or necrotic pulp. Clinical success will be defined by the absence of pain, swelling, sinus tract, mobility, or tenderness to percussion. Radiographic success will be defined by the absence of periapical or inter-radicular radiolucency, internal or external resorption, and evidence of continued root resorption consistent with normal exfoliation.

SECONDARY OUTCOMES:
Anxiety Level using RMS Pictorial Scale | Baseline (in the waiting area before entering the operatory), Pre-operative (immediately before the start of the procedure), Operative (during the dental treatment), and Post-operative (immediately after completion of the procedure).
  Anxiety will be assessed using the Raghavendra Madhuri Sujata (RMS) Pictorial Scale, a validated visual scale designed to measure dental anxiety in children. Scores range from 1 to 5, where a higher score indicates a greater level of anxiety.
Pulse Rate in beats per minute (bpm) using Pulse Oximeter | Baseline (in the waiting area before entering the operatory), Pre-operative (immediately before the start of the procedure), Operative (during the dental treatment), and Post-operative (immediately after completion of the procedure).
  Pulse rate will be measured in beats per minute (bpm) using a calibrated digital pulse oximeter to assess the physiological response to anxiety during dental treatment.
Oxygen Saturation (SpO₂) in percentage (%) using Pulse Oximeter | Baseline (in the waiting area before entering the operatory), Pre-operative (immediately before the start of the procedure), Operative (during the dental treatment), and Post-operative (immediately after completion of the procedure).
  Oxygen saturation (SpO₂) will be measured in percentage (%) using a calibrated digital pulse oximeter to assess physiological changes associated with anxiety during dental treatment.